CLINICAL TRIAL: NCT02670499
Title: A Randomized Controlled Multicenter Study Comparing GAP-FLEX to Continuous Passive Motion (CPM) Therapy in Combination With Standard of Care Physical Therapy in Subjects With Total Knee Replacement (TKR)
Brief Title: Study Comparing GAP-Flex to CPM Therapy in Treatment of TKR
Acronym: GAP-Flex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xeras Medical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GPF2015-01
Record Dates: First submitted 2015-09-04; First posted 2016-02-01 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Total Knee Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GAP-FLEX (Experimental): Study Device will be used up to 6 times per day for up to 6 minutes to aid in the recovery and improve the degree of flexion from TKR
  Interventions: Device: GAPFLEX
- CPM (Active Comparator): Control Device will be used up to 2 hours per day for up to 3 times per day to aid in the recovery and improve the degree of flexion from TKR and be compared to the Study Device
  Interventions: Device: CPM

INTERVENTIONS:
Device: CPM — Used to aid in recovery from TKR
  Other Names: Continuous Passive Motion Device
  Arms: CPM
Device: GAPFLEX — Used to aid in the recovery of TKR
  Arms: GAP-FLEX

SUMMARY:
Post Market TKR study

DETAILED DESCRIPTION:
A post-market study to evaluate the safety and effectiveness of the GAP-FLEX device in combination with standard of care physical therapy compared to the standard of care CPM device in combination with standard of care physical therapy in Subjects who have undergone TKR

ELIGIBILITY:
Inclusion Criteria:

* Minimum age 50 years
* Subject is undergoing total knee replacement
* Subject agrees to comply with the physical therapy regime

Exclusion Criteria:

* With a flexure contracture > 10 degrees
* Degree of flexion < 60 degrees pre-procedure or immediately post-procedure
* Severe motion restriction as determined by the investigator
* Severe deformity determined by the investigator
* Taking chronic pain medication for use other than knee pain
* Post surgery hospital stay is > 4 days
* Knee disorders other than osteoarthritis
* With fibromyalgia
* Chronic narcotic use as determined by the investigator.
* Have a medical or psychological history that in the opinion of the investigator would make the subject a poor candidate for the study.
* Who need a revision implant
* Who have participated in clinical study within the past 30 days (prior to enrollment) that may affect the outcome of this study
* Amputations below or above knee of non-operated leg
* Weight is >250 pounds and/or morbidly obese (BMI > 40)
* History of blood clots
* Deep vein thrombosis
* Females who are pregnant
* Females who wish to become pregnant during the length of study participation
* Subjects with any of the following post-surgery conditions;
* Screws needed
* Intraoperative identification of a fracture or soft bone
* Admitted to ICU
* Additional procedures (other than TKR) needed for other identified or pre-existing conditions

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-11-18 (Actual); Primary Completion 2017-02-07 (Actual); Study Completion 2017-06-23 (Actual)

PRIMARY OUTCOMES:
Flexion | Degree of flexion achieved at week 4 visit
  improvement in week 4 visit degree of flexion measured by Goniometer in the GAP-FLEX group will be compared to the CPM

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Nix Orthopaedic Center, San Antonio, Texas
  - Orthopaedic Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No